CLINICAL TRIAL: NCT02048839
Title: Long-term Effects of Lifestyle Intervention During Pregnancy in High Risk Women and in Their Offspring - Role of Environmental, Genetic and Epigenetic Factors
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Saila Koivusalo, MD PhD, Helsinki University Central Hospital
Other Study IDs: Radiel 5Y
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, hair, urine and fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Radiel Intervention group and their children: Participated the Radiel- intervention study (2008-2011) in the Intervention group: Lifestyle counselling during and after pregnancy (up to 1 year post partum)
- Radiel Control Group with their children: Control group in the Radiel- intervention study.

SUMMARY:
SUBJECTS:

All participants in the RADIEL-study (2008-2011) who delivered (n=535), will be invited to this follow-up study, with their children (age 3-5 years) and the father. The investigations are carried out during two separate visits. The father receives mail questionnaires

OVERALL OBJECTIVES:

1. To determine the long-term effectiveness of a lifestyle intervention in high risk women and their offspring a in reducing the incidence of T2DM and cardiovascular disease and their risk factors b in preventing obesity c on biomarkers d on genetic and epigenetics markers .
2. To study the association between maternal diet during pregnancy and metabolic markers in the offspring at age 3-5 years.
3. To study the association between maternal exercise habits during pregnancy and metabolic markers in the offspring at age 3-5 years.
4. To study the association between maternal a) glucose-insulin metabolism b) lipid metabolism c) adipoinsulinar axis and d) inflammatory markers and birth size and later health outcomes in the mothers and their offspring.
5. To study the association between gut microbiota and markers of offspring health
6. To study associations between offspring cardiovascular morphology/function, offspring body size/composition, and maternal cardiovascular risk
7. To study the cost effectiveness of the intervention.

METHODS:

Maternal measurements

1. Height, weight, waist and hip circumference
2. Blood pressure, pulse
3. Body fat percentage
4. Blood tests e.g. markers of glucose metabolism and lipids, vitamin D, Calcium and bone markers, DNA sample and inflammation markers
5. Fecal and hair samples
6. Diurnal salivary cortisol assessment
7. Background questionnaire: socioeconomic and health-related background
8. Health-related quality of life (15-D).
9. 3-day food diary and exercise diary
10. ArmBand (acceleration sensor), assessment of physical activity and sleep for 7 days
11. Psychological questionnaires
12. Pulse wave velocity (PWV) will be assessed
13. Advanced glycation endproducts - a marker of cardiovascular health will be assessed
14. Dental and oral health
15. Bone health
16. VHRU of arterial structure

Paternal measurements

1. Background questionnaire (incl. height, weight, age)
2. DNA-sample (buccal)
3. 3-day food diary
4. Psychological questionnaires
5. Physical activity questionnaire (12 months)

Measurements of children

1. Body weight, height, blood pressure, pulse
2. Body fat percentage
3. Psychological questionnaires
4. Food and physical activities diaries
5. ActiGraph, assessment of physical activity and sleep for 7 days
6. Blood samples e.g. glucose- and insulin metabolism, lipids, vitamin D and calcium metabolism, DNA-sample and samples for inflammation markers
7. Fecal, urine and hair samples
8. A copy of child welfare center card (e.g. data on growth, immunizations, health)
9. Endothelial function and pulse wave velocity (PWV)
10. Bone health with peripheral CT
11. Heart structure and function
12. VHRU of arterial structure

TIMETABLE

Follow up starts in January 2014, and will continue until 2018. Data analysis starts in 2017 and results will be reported from 2018 onwards in international peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* all study subjects form Radiel intervention study, who delivered a baby

Exclusion Criteria:

* none.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women who participated the Radiel intervention study, and were originally randomly assigned to either active lifestyle intervention group or control group. They were all high risk women with BMI >30 or prior gestational GDM. To this follow up-study we invite also the children born during the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 680 (Actual)
Dates: Start 2014-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Type 2 Diabetes | 3-5 years post partum

SECONDARY OUTCOMES:
Metabolic syndrome and cardiovascular morbidity | 3-5 years post partum

OTHER OUTCOMES:
Obesity | 3-5 years post partum

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University, Helsinki, Finland